CLINICAL TRIAL: NCT07332052
Title: Comparison of Parameters That Can be Used to Predict Frailty in Elderly Femur Fracture Patients.
Brief Title: Predicting of Frailty
Acronym: PRE-FRAIL
Status: Not yet recruiting | Type: Observational
Sponsor: ali ihsan uysal (Other)
Responsible Party: Sponsor-Investigator, ali ihsan uysal, Ass.Prof., Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Other Study IDs: 250066
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Femur Fractures; Frailty; Sarcopenia
Keywords: Geriatric Anesthesia; Frailty; Hip Fracture; Sarcopenia; Rectus Femoris
MeSH Terms: conditions — Femoral Fractures; Frailty; Sarcopenia; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly Hip Fracture Patients: Patients aged 65 and older who have been diagnosed with a trochanteric femur fracture and are scheduled for orthopedic surgery.
  Interventions: Other: Clinical and Functional Assessment; Other: Rectus femoris thickness measurement

INTERVENTIONS:
Other: Clinical and Functional Assessment — Assessment of frailty status using the Clinical Frailty Scale and measurement of handgrip strength using a hand dynamometer (measured in kilograms). Ultrasonographic measurement of the rectus femoris muscle thickness (mm) and femur-skin distance (mm) conducted one day before surgery.
  Other Names: Clinical Frailty Scale; Hand Dynamometry; Rectus Femoris Ultrasound; Sarcopenia Screening via Ultrasound
Other: Rectus femoris thickness measurement — By using ultrasound linear prob the thickness of rectus femoris muscle will be measured

SUMMARY:
This study aims to evaluate the frailty status of elderly patients undergoing surgery for hip fractures (femur trochanteric fractures). Since frailty is a critical factor in surgical outcomes and recovery, researchers want to find simple, fast, and objective ways to measure it. This study will investigate muscle thickness measured by ultrasound, handgrip strength measured by a dynamometer, and routine blood test values can accurately predict a patient's frailty level. If these objective methods are proven effective, it will help anesthesia and surgical teams manage the perioperative process more safely for high-risk elderly patients

DETAILED DESCRIPTION:
65 and over years old elderly patients admitted to the orthopedics department with a diagnosis of trochanteric femur fracture will be enrolled in this study.

Preoperative Assessment: A researcher anesthesiologist, who is not involved in the patient's perioperative clinical management, will conduct the assessments to ensure objectivity. One day prior to the scheduled surgery, the following procedures will be performed:

Frailty Evaluation: Clinical frailty status will be determined using the Clinical Frailty Scale. In conjunction with this, handgrip strength will be measured using a calibrated hand dynamometer.

Ultrasonographic Measurements: Ultrasound will be used to measure the thickness of the rectus femoris muscle and the distance from the femur to the skin. These measurements will serve as objective indicators of musculoskeletal status.

Data Collection: Demographic data (age, weight, height, comorbidities) and routine preoperative laboratory results will be recorded from the hospital's electronic medical records. Laboratory parameters to be analyzed include:

Hematological: Hemoglobin, MPV, MCV, Neutrophil, and Lymphocyte counts.

Biochemical: Albumin, Creatinine, CRP, and GFR.

The study focuses on evaluating the correlation between these objective measurements (ultrasound and dynamometry) and the established clinical frailty scores to determine their predictive value in the geriatric surgical population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older.
* Confirmed diagnosis of trochanteric femur fracture.
* Planned for orthopedic surgery under general or regional anesthesia.
* Ability to provide written informed consent (either by the patient or a legal representative).

Exclusion Criteria:

* Patients with advanced dementia or severe cognitive impairment who cannot cooperate with the handgrip strength test or Fried criteria questionnaire.
* Patients with terminal-stage diseases or those under palliative care.
* History of neuromuscular diseases or severe muscle-wasting conditions that affect the lower limbs (e.g., advanced muscular dystrophy).
* Patients with active infections or skin lesions at the site of ultrasound measurement (rectus femoris area).
* Emergency cases requiring immediate surgery where preoperative assessment cannot be completed.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population consists of geriatric patients aged 65 years and older who have been hospitalized at the Orthopedics and Traumatology department of Mugla Sitki Kocman University Training and Research Hospital with a diagnosis of trochanteric femur fracture. This population includes patients scheduled for elective or semi-urgent orthopedic surgery who are capable of undergoing preoperative clinical and ultrasonographic assessments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Correlation between Rectus Femoris Muscle Thickness and Frailty Score | Preoperative (within 24 hours before surgery)
  Evaluation of the relationship between clinical frailty status (measured by the Clinical Frailty Scale) and objective muscle mass (measured as rectus femoris thickness in millimeters via ultrasonography). Over 5 point indicate frailty.

SECONDARY OUTCOMES:
Predictive Value of Handgrip Strength for Frailty | Preoperative
  Assessment of handgrip strength using a hand dynamometer to evaluate its correlation with the Frailty Score.
Correlation of Laboratory Biomarkers with Frailty Status | 1 day before operation
  Evaluation of the relationship between frailty and preoperative blood levels of Albumin, C-Reactive Protein (CRP), Glomerular Filtration Rate (GFR)
Hematological Indicators of Frailty | 1 day before operation
  Analysis of Hemoglobin levels and Neutrophil-to-Lymphocyte Ratio (NLR) in relation to the patient's frailty score.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University Training and Research Hospital, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect the privacy of the participants and to maintain confidentiality in accordance with the institutional review board's (Mugla Sitki Kocman University Ethics Committee) regulations and local data protection laws.

REFERENCES:
- [Result] Mehmet H, Yang AWH, Robinson SR. Measurement of hand grip strength in the elderly: A scoping review with recommendations. J Bodyw Mov Ther. 2020 Jan;24(1):235-243. doi: 10.1016/j.jbmt.2019.05.029. Epub 2019 May 24. PMID 31987550
- [Result] Sabatino A, Regolisti G, Bozzoli L, Fani F, Antoniotti R, Maggiore U, Fiaccadori E. Reliability of bedside ultrasound for measurement of quadriceps muscle thickness in critically ill patients with acute kidney injury. Clin Nutr. 2017 Dec;36(6):1710-1715. doi: 10.1016/j.clnu.2016.09.029. Epub 2016 Oct 1. PMID 27743614
- [Result] Saglam Oz M, Toprak B, Bora R, Demir I. The Role of Hematological Parameters in Critically Ill Patients: Mortality Prediction in Elderly Intensive Care Unit Patients. Cureus. 2025 Apr 13;17(4):e82183. doi: 10.7759/cureus.82183. eCollection 2025 Apr. PMID 40364870